CLINICAL TRIAL: NCT06023641
Title: A Protocol for the Treatment of Newly Diagnosed Rhabdomyosarcoma Using Molecular Risk Stratification and Liposomal Irinotecan Based Therapy in Children With Intermediate and High Risk Disease
Brief Title: Treatment of Newly Diagnosed Rhabdomyosarcoma Using Molecular Risk Stratification and Liposomal Irinotecan Based Therapy in Children With Intermediate and High Risk Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMS2021; NCI-2024-00701 (Other: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2023-08-27; First posted 2023-09-05 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Rhabdomyosarcoma
MeSH Terms: conditions — Rhabdomyosarcoma | interventions — Vincristine; Dactinomycin; Cyclophosphamide; Brachytherapy; irinotecan sucrosofate; Vinorelbine; Temozolomide; Filgrastim; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Low -risk (Experimental): The participant will receive 12 weeks (4 cycles) of VAC chemotherapy (vincristine, dactinomycin and cyclophosphamide) followed by 12 weeks (4 cycles) of VA chemotherapy (vincristine, dactinomycin).
  Each cycle of VAC/VA chemotherapy will last for 3 weeks, for a total of 12 weeks (VAC or VA will be given in Week 1 of each cycle and vincristine will be given Weeks 2 and 3). At week 12, the participant will have scans and tests to reevaluate your tumor's response to the treatment. After surgery and radiation, the participant will receive an additional 12 weeks (4 cycles) of the same chemotherapy without cyclophosphamide. Vincristine and dactinomycin, also called "VA". After 4 cycles of VA, The investigator will re-evaluate the tumor again at week 24 and the patient will not get any more chemotherapy, but will be closely watched for any signs of tumor recurrence.
  Interventions: Drug: Vincristine; Drug: Dactinomycin; Drug: Cyclophosphamide; Procedure: Surgical Resection; Procedure: Proton beam radiation or external beam radiation or brachytherapy
- Intermediate-risk (Experimental): The purpose of this part of the study is to find out if adding a drug called liposomal irinotecan (also called Onivyde) to standard chemotherapy/radiation/surgery will result in better treatment outcomes for patients with intermediate and high risk rhabdomyosarcoma. The investigators also want to find the best radiation dose to give for intermediate and high risk patients who have large tumors (> 5 cm).
  The patient will receive 42 weeks of VAC chemotherapy (vincristine, actinomycin D/dactinomycin and cyclophosphamide) alternating with VLI chemotherapy (vincristine/liposomal irinotecan). The participant will also have surgery to remove the tumor and radiation therapy during this time. After this therapy is completed you will get an additional 6 months of maintenance chemotherapy with vinorelbine and oral (by mouth) cyclophosphamide.
  Interventions: Drug: Vincristine; Drug: Dactinomycin; Drug: Cyclophosphamide; Procedure: Surgical Resection; Procedure: Proton beam radiation or external beam radiation or brachytherapy; Drug: Liposomal irinotecan; Drug: Vinorelbine; Drug: Filgrastim, peg-filgrastim
- High-risk (Experimental): The purpose of this part of the study is to find out if adding a drug called liposomal irinotecan (also called Onivyde) to standard chemotherapy/radiation/surgery will result in better treatment outcomes for patients with high risk rhabdomyosarcoma. The investigator also want to find the best radiation dose to give for high risk patients who have large tumors (> 5 cm).
  The patient will receive 42 weeks of VAC chemotherapy (vincristine, actinomycin D/dactinomycin and cyclophosphamide) alternating with VLIT chemotherapy (vincristine/liposomal irinotecan/temozolomide). Also having surgery to remove the participants tumor and radiation therapy during this time. After this therapy is completed the patient will get an additional 6 months of maintenance chemotherapy with vinorelbine and oral (by mouth) cyclophosphamide.
  Interventions: Drug: Vincristine; Drug: Dactinomycin; Drug: Cyclophosphamide; Procedure: Surgical Resection; Procedure: Proton beam radiation or external beam radiation or brachytherapy; Drug: Liposomal irinotecan; Drug: Vinorelbine; Drug: Temozolomide; Drug: Filgrastim, peg-filgrastim

INTERVENTIONS:
Drug: Vincristine — Low -risk Administer IV push over 1 minute (or infusion via minibag as per institutional standards) on Day 1 of Weeks 1,8, 15 (3) doses. The maximum dose is 2 mg for all participants.
  Intermediate-risk Administer IV, over 1 minute, 3 doses, weekly on day1 High-risk Administer by IV infusion over 1 minute, 3 doses, weekly on day 1,8,15
  Other Names: Oncovin
Drug: Dactinomycin — Low-risk Administer by slow IV push over 1-5 minutes on Day 1 of Weeks 1, (1) dose. The maximum dose is 2.5 mg for all participants.
  Intermediate-risk Administer by slow IV over 1-5 minutes., 1 doses weekly on day 1 High-risk Administer by slow IV over 1-5 minutes, day1
  Other Names: (actinomycin-D)
Drug: Cyclophosphamide — Low-risk Administer by IV infusion over 30-60 minutes on Day 1, 91) dose, Mesna and hydration will be given with IV cyclophosphamide according to institutional standards.
  Intermediate-risk Administer by IV infusion over 30-60 minutes, 1 dose, day 1 High-risk Administer by IV infusion over 30-60 minutes, 1 dose, day1
  Other Names: Cytoxan®.
Procedure: Surgical Resection — Low, Intermediate and High-risk
Procedure: Proton beam radiation or external beam radiation or brachytherapy — Low, Intermediate and High-risk
Drug: Liposomal irinotecan — Intermediate and High-risk Administer by IV infusion over 90 minutes, 1 dose on day 1 Liposomal irinotecan should be premedicated with dexamethasone (or an equivalent corticosteroid) if not contraindicated. Premedication with diphenhydramine and an H2 receptor antagonist (i.e., famotidine) are also encouraged.
  Other Names: (Onivyde®)
  Arms: High-risk; Intermediate-risk
Drug: Vinorelbine — Intermediate and High-risk Administer via slow IV push over 6-10 minutes (or infusion via minibag as per institutional standards) on Day 1 of Weeks 43-45, 47-49, 51-53, 55-57, 59-61, 63-65.
  Other Names: Navelbine
  Arms: High-risk; Intermediate-risk
Drug: Temozolomide — High-risk Administer PO (or by NG or G tube) 5 doses, on Days 1-5 When administering with liposomal irinotecan, administer temozolomide prior to liposomal irinotecan. Preferably, administer on an empty stomach (at least 1 hour before and 2 hours after food) to improve absorption. When using temozolomide capsules, round dose to the nearest 5 mg capsule. The capsule may be opened, and contents mixed with applesauce or apple juice. A compounded oral suspension is also available. If emesis occurs within 20 minutes of taking a dose of temozolomide, then the dose may be repeated once.
  Other Names: Temodar
  Arms: High-risk
Drug: Filgrastim, peg-filgrastim — Low, Intermediate and High-risk:
  Prophylactic myeloid growth factor support (Filgrastim or Pegfilgrastim) should be used after all VAC cycles for patients on the high-risk arm. Start myeloid growth factor support (for example, filgrastim 5 mcg/kg/dose SubQ daily until the ANC is ≥ 2000/μL after the expected nadir OR pegfilgrastim 0.1 mg/kg/dose [for patients < 45 kg] or 6 mg/dose [for patients ≥ 45 kg] SubQ x 1 dose) 24-48 hours after VAC cycles. Filgrastim may be continued without regard to VCR. Discontinue filgrastim at least 24 hours before the start of the next cycle. Prophylactic myeloid growth factor support should NOT be used after VLIT cycles or during maintenance chemotherapy.
  Other Names: Neupogen
  Arms: High-risk; Intermediate-risk

SUMMARY:
This is a phase II study to determine safety and efficacy of combining liposomal irinotecan with vincristine alternating with VAC in intermediate-risk patients, liposomal irinotecan with temozolomide and vincristine alternating with VAC in high-risk patients and the chemotherapy combinations when given with concomitant radiation therapy in intermediate and high risk patients.

Primary Objective

* Estimate event-free survival for intermediate-risk participants treated with VAC and vincristine and liposomal irinotecan (VLI) with the addition of maintenance therapy with vinorelbine and cyclophosphamide.
* Estimate the event-free survival for high-risk patients treated with VAC and vincristine, liposomal irinotecan, and temozolomide with the addition of maintenance therapy with vinorelbine and cyclophosphamide.

Secondary Objectives

* To assess the relation between pharmacogenetic variation in CEP72 genotype and vinca alkaloid (vincristine; vinorelbine) disposition in children with rhabdomyosarcoma.
* To assess the relation between the pharmacogenetic variation in drug metabolizing enzymes and drug transporters, and the pharmacokinetics of vinca alkaloids, liposomal irinotecan, and cyclophosphamide in children with rhabdomyosarcoma.
* To assess the extent of inter-patient variability in the pharmacokinetics of vinca alkaloids, liposomal irinotecan, and cyclophosphamide in children with rhabdomyosarcoma, and explore possible associations between drug disposition and patient specific covariates (e.g., age, sex, race, weight).
* Estimate the cumulative incidence of local recurrence and overall 3-year event-free survival in patients with low-risk disease, intermediate-risk disease or high-risk disease treated with either no adjuvant radiation or minimal volume radiation and compare these outcomes with the outcomes achieved on RMS13.

DETAILED DESCRIPTION:
This is a phase II study to determine safety and efficacy of combining liposomal irinotecan with vincristine alternating with VAC in intermediate-risk patients, liposomal irinotecan with temozolomide and vincristine alternating with VAC in high-risk patients and the chemotherapy combinations when given with concomitant radiation therapy in intermediate and high risk patients. The dose of liposomal irinotecan for intermediate and high risk patients will be 160/mg/m2 on Day 1 based on the results and recommended phase 2 dose of the Phase I trial ONITT trial. The primary objective is to assess event-free survival (EFS). The sample size is determined based on a 2-year EFS estimate for each risk group, with a total study duration of 4 years for enrollment and 2 years of follow-up per patient.

The study employs a single-arm adaptive Phase II design, with an estimated 46 patients in the intermediate-risk group and 34 patients in the high-risk group, ensuring 80% power and a 5% Type I error rate. The trial will conclude once the last enrolled patient has completed 2 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

• Newly diagnosed participants with the diagnosis of rhabdomyosarcoma (RMS) of any subtype. This includes embryonal rhabdomyosarcoma (fusion negative), alveolar rhabdomyosarcoma (fusion positive), as well as spindle cell and sclerosing

• Must have either low-, intermediate-risk or high-risk disease, defined as:

1. Low-risk: TP53 and MYOD1 negative AND

   • Embryonal, congenital/infantile spindle cell, or spindle cell/sclerosing FOXO1 fusion negative histology
   * Stage 1 Group I, Group II
   * Stage 1 Group III orbital only
   * Stage 2 Group I, Group II
2. Intermediate-risk: MYOD1 and TP53 negative AND

   • Embryonal, congenital/infantile spindle cell, or spindle cell/sclerosing FOXO1 fusion negative histology o Stage 1 Group III non orbit o Stage 3 Group I/II

   o Stage 2/3 Group III
   * Stage 4 Group IV and Oberlin 0-1

     • Alveolar, spindle cell/sclerosing FOXO1 fusion positive histology
   * Stage 1-3, Group I-III N0
3. High-risk: All MYOD1 and TP53 mutant tumors regardless of stage and Group AND/OR

   * Embryonal, congenital/infantile spindle cell or spindle cell/sclerosing FOXO1 fusion negative o Group IV ≥ 10 year of age and Oberlin ≥ 2
   * Alveolar, spindle cell/sclerosing FOXO1 fusion positive

     * N1
     * Stage 4 Group IV

   See Appendices I and II for Staging and Clinical Grouping.

   Age < 22 years (eligible for enrollment until 22nd birthday)

   • Performance level corresponding to ECOG score of 0, 1, or 2. The Lansky performance score should be used for participants < 16 years (see Appendix VII).
   * Participant has received no prior radiotherapy or chemotherapy for rhabdomyosarcoma (excluding steroids) unless an emergency situation requires local tumor treatment (discuss with PI).
   * Initiation of chemotherapy is planned within 6 weeks (42 days) of the definitive biopsy or surgical resection.
   * Adequate bone marrow function defined as:
   * Peripheral absolute neutrophil count (ANC) ≥ 750/μL
   * Platelet count ≥ 75,000/μL (transfusion independent)
   * Adequate liver function defined as total bilirubin < 1.5 x upper limit of normal (ULN) for age. Participants with biliary or hepatic primaries with bilirubin values greater than 1.5 x ULN may be enrolled on study if all other eligibility criteria are met.

   Adequate renal function defined as:

   Creatinine clearance or radioisotope GFR > 70 mL/min/1.732 or serum creatinine based on age as follows:

   Age Maximum serum creatinine (mg/dL) Male Female

   1 month to < 6 months 0.4 0.4 6 months to < 1 year 0.5 0.5 Age Maximum serum creatinine (mg/dL)
   1. to < 2 years 0.6 0.6
   2. to < 6 years 0.8 0.8

   6 to < 10 years 1 1 10 to < 13 years 1.2 1.2 13 to < 16 years 1.5 1.4 > 16 years 1.7 1.4

   The threshold creatinine values in this table were derived from the Schwartz formula for estimating GFR25 utilizing child length and stature. Data published by the CDC.

   Participants with urinary tract obstruction by tumor must meet the renal function criteria listed above AND must have unimpeded urinary flow established via decompression of the obstructed portion of the urinary tract.

   • Adequate pulmonary function defined as: no evidence of dyspnea at rest and a pulse oximetry > 94% if there is a clinical indication for determination. Pulmonary function tests are not required.

   • Patients requiring emergency radiation therapy are eligible for enrollment on this trial. See Section 4.11 for radiation therapy guidelines.

   • No evidence of active, uncontrolled infection.

   All participants and/or their parents or legal guardians must sign a written informed consent.

   Exclusion Criteria:

   • Patients who have received any chemotherapy (excluding steroids).

   • Patients who have received prior full course RT at the primary site of disease. This does not exclude patients that received emergent radiation.
   * Ongoing or history of non-infectious interstitial lung disease requiring significant medical intervention.
   * Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation and for at least 3 months after treatment is completed.
   * Female patients who are pregnant are not eligible since fetal toxicities or teratogenic effects have been noted for several of the study drugs. Female participants > 10 years of age or post-menarchal must have a negative serum or urine pregnancy test within 24 hours prior to beginning treatment.
   * Lactating females who are or plan to breastfeed their infants are not eligible.

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 135 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2034-10 (Estimated); Study Completion 2037-10 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated doses (MTDs) | 4 years
  MTD is defined in the study as the highest treatment dose that would deliver desirable treatment effects without resulting in a target toxicity rate greater than 0.3. For each of three groups (intermediate-risk, high-risk, and intermediate-and-high-risk-with-early-radiation), we will employ the Bayesian optimal interval (BOIN) design to find the MTD.
Event-free survival (EFS) | 2 years post, off therapy
  We will estimate the 2-year event-free survival for intermediate-risk and high-risk patients, which is the estimated probability of a patient not having any events within the 2-year follow-up. If an event, including local failure, distant failure, death or loss to follow-up occurs for a patient within 2-year, we call it failure, otherwise call it response.
Local recurrence rate (LRR) | 2 years
  LRR is defined as a binary endpoint in the study. The local recurrence-free survival (LRFS) is defined as time from randomization to the earlier date of the first of local disease recurrence or death due to any cause. The distant failure will be considered to be the competing risk, patients for whom follow-up ended without clinical improvement will be censored. The goal of the local recurrence rate endpoint is to evaluate the 2-year LRR by comparing the administration of 59.4 GyRBE and 68 GyRBE for patients (pooled intermediate- and high-risk groups) with tumor size greater than or equal to 5cm meeting the eligibility criteria for randomization (no biliary tree or specific extremity cases).
  .

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Pappo, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (3):
- United States (3):
  - Stanford University, Palo Alto, California
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols